CLINICAL TRIAL: NCT01741480
Title: Comparing an Early Warning Alert With a Standardized Triage Intervention to Standard Care for the Management of Hospitalized Patients on General Hospital Wards.
Brief Title: Early Warning System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other); American College of Chest Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201210003
Record Dates: First submitted 2012-11-27; First posted 2012-12-05 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Congestive Heart Failure; Chronic Obstructive Pulmonary Disease; Cancer; Diabetes Mellitus; Obstructive Sleep Apnea
Keywords: Outcomes; Early warning systems; ICU transfer
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Neoplasms; Diabetes Mellitus; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine care (Placebo Comparator): General hospital ward patients will receive routine care.
  Interventions: Other: routine care
- Intervention arm (Experimental): The intervention with early warning system monitoring is to have the rapid response team assess the patients real-time.
  Interventions: Other: Early warning system monitoring.

INTERVENTIONS:
Other: Early warning system monitoring. — General hospital ward patients will be monitored 24/7 for clinical deterioration using the early warning system monitoring developed at Washington University.
  Arms: Intervention arm
Other: routine care
  Arms: Routine care

SUMMARY:
The study will begin in 2013 whereby patients having an early warning system (EWS) alert will be randomized to be seen by the rapid response team (RRT) for triage versus usual care. A RRT is usually made up of a nurse and/or a physician who respond to a requested activation of the RRT (called an "ACT"). The intervention will occur as follows:

DETAILED DESCRIPTION:
The study will begin in 2013 whereby patients having an early warning system (EWS) alert will be randomized to be seen by the rapid response team (RRT) for triage versus usual care. A RRT is usually made up of a nurse and/or a physician who respond to a requested activation of the RRT (called an "ACT"). The intervention will occur as follows:

1. Real-time monitoring of the eight general hospital wards (GHWs)((10100, 10200, 11100,11200, 12100, 12200, 14400, 14500)will occur 24 hours daily. Through multiple past collaborative efforts and studies involving interventions at BJH, informatics personnel have already demonstrated that they can accomplish this task using their computing and algorithmic resources. The prediction tool (PT) employed is a validated PT aimed at identifying any form of clinical deterioration occurring on a GHW requiring ICU transfer or leading to patient death.
2. Patients meeting the prediction criteria for an increased risk of clinical deterioration will be identified on the GHWs. An automated text message will be generated that provides the patient's name, their room number, the date and time of the message, and text indicating that they meet the criteria for risk of deterioration. Messages will only be generated for patients assigned to the intervention group.
3. The EWS text message will be sent to the on-call RRT nurse's phone. These are phones that are transferred from one RRT nurse to the other as changes of shift occur. It is their primary means of communicating with the hospital.
4. The RRT nurse for the intervention patients will go into the flagged patient's room within 10 to 15 minutes of receiving the message and perform a clinical assessment. Based on the RRT nurse's assessment either no additional action need occur or he/she will call either the physician on duty or activate an ACT as well as apply the "four D's", which was internally established at Barnes-Jewish Hospital (BJH) for treatment of patients on GHWs identified to have impending clinical deterioration. The four "D's" refer to the following: Discuss level of care, Drugs for treatment (e.g., antibiotics), Diagnostics (lab tests, cultures), and Damage control (e.g., use of intravenous fluids, oxygen).

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized on the General Hospitals Wards of Barnes-Jewish Hospital.

Exclusion Criteria:

* Patients with a do-not-resuscitate order,
* Patients not expected to survive their hospitalization.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marin Kollef, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Routine Care: General hospital ward patients will receive routine care.
  routine care =286
- Intervention Arm: Patients will have active surveillance by the early warning system performed on a real-time basis to identify clinical deterioration.
  Early warning system monitoring.: General hospital ward patients will be monitored 24/7 for clinical deterioration using the early warning system developed at Washington University. = 285
Period: Overall Study
Arm/Group | Routine Care | Intervention Arm
Started | 285 | 286
Completed | 285 | 286
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Routine Care: General hospital ward patients will receive routine care.
  routine care
- Intervention Arm: Patients will have active surveillance by the early warning system performed on a real-time basis to identify clinical deterioration.
  Early warning system monitoring.: General hospital ward patients will be monitored 24/7 for clinical deterioration using the early warning system developed at Washington University.
- Total: Total of all reporting groups
Arm/Group | Routine Care | Intervention Arm | Total
Number analyzed (Participants) | 285 | 286 | 571
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (15.4) | 63.7 (16) | 63.3 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 132 | 272
  Male | 145 | 154 | 299
Region of Enrollment [Number; unit: participants] — Saint louis Region
  participants
    United States | 285 | 286 | 571

OUTCOME MEASURES:

1. Primary Outcome: ICU Transfer
Description: Patients transferred to the ICU from a general hospital ward will be assessed as having met the outcome.
Time Frame: Patients will be assessed for the primary outcome measure during their hospital with an average of 14 days.
Measure: Number; unit: participants
Arm/Group | Routine Care | Intervention Arm
Number analyzed (Participants) | 285 | 286
participants | 52 | 51

2. Secondary Outcome: Mortality
Description: Death during hospitalization will be used to determine the presence of this outcome.
Time Frame: Patients will be asessed for the secondary outcome measure during an average of 28 days..
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Routine Care | Intervention Arm
Serious Adverse Events (participants affected / at risk) | 0/285 | 0/286
Other Adverse Events (participants affected / at risk) | 0/285 | 0/286

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No